CLINICAL TRIAL: NCT06674044
Title: Effect of SLC01B1 (rs2306283) Polymorphism on the Efficacy and Safety Profile of Atorvastatin in Pakistani Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Riphah/IIMC/IRC/23/30104
Record Dates: First submitted 2024-09-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood was withdrawn, and DNA extraction was performed using Chelex method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Atorvastatin — Atorvastatin 10mg once a day for 1 month

SUMMARY:
The goal of this prospective cohort study was to identify the effect of SLC01B1 gene polymorphism in the Pakistani population. The main questions it aims to answer are:

To identify polymorphism in SLOC1B1 (rs2306283) in the Pakistani population. To determine the association between SLOC1B1 (rs2306283) polymorphism and the clinical efficacy of atorvastatin To determine the association between SLOC1B1 (rs2306283) polymorphism and the safety profile of atorvastatin.

DETAILED DESCRIPTION:
The goal of this prospective cohort study was to identify the effect of SLC01B1 gene polymorphism in the Pakistani population, due to the high prevalence of this variant in the Pakistani Population

The main questions it aims to answer are:

To identify polymorphism in SLOC1B1 (rs2306283) in the Pakistani population. To determine the association between SLOC1B1 (rs2306283) polymorphism and the clinical efficacy of atorvastatin To determine the association between SLOC1B1 (rs2306283) polymorphism and the safety profile of atorvastatin.

The participants' blood samples were taken and further genotyping was performed using conventional tetraARMS PCR. The results were visualized by gel electrophoresis.

ELIGIBILITY:
Inclusion Criteria:

1. Pakistani individuals aged between 30 to 60 years
2. Patients with deranged lipid profile
3. Newly diagnosed patients of dyslipidemia taking atorvastatin (Lipiget) 10mg/day
4. Normal hepatic and renal function

Exclusion Criteria:

1. Patient taking other lipid-lowering medications
2. Moderate and severe systemic diseases
3. Pregnancy
4. Patients taking medications and diet that can interact with atorvastatin
5. Hypothyroidism
6. Recent history of surgical procedure or trauma

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pakistani Population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
To identify genetic polymorphism in SLOC1B1 in the Pakistani population | 1 month
  Genetic polymorphism in SLOC1B1 in the Pakistani population will be assessed by ARMS PCR assay.
Lipid profile | 1 month
  Lipid profile will be measured at 0 and on the 28th day of atorvastatin therapy on a blood sample.
  LDL cholesterol was categorized as optimal <100mg/dl, Near or above optimal = 100-129mg/dl, Borderline = 130-159mg/dl, high = 160-189mg/dl, and very high >190mg/dl.
  Total cholesterol: <200mg/dl = desirable, 200-239mg/dl = borderline high, >240mg/dl = high.
  HDL cholesterol: <40mg/dl = low and >60mg/dl = high.
  Triglycerides: <150mg/dl were considered optimal, 150-199mg/dl as Borderline high, and 200-500 mg/dl as high
The SAMS-CI tool | 1 month
  The patient will be assessed for safety profile through the myopathy by Statin-associated myopathy (SAM-CI) tool by filling out the questionnaire on days 0, 14, and 28. The SAMS-CI tool will be used, to record the location, symmetry, and onset of muscle symptoms at day 0, 14, and 28 of atorvastatin therapy. Patients reporting the presence of muscular pain will be further divided into "Unlikely", "Possible", and "Probable" categories based on their SAMS-CI score.

CONTACTS AND LOCATIONS:
Overall Officials: Tayaba Farooq, MBBS, Principal Investigator — Riphah International University
Locations (1):
- IIMC, Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hedayatnia M, Asadi Z, Zare-Feyzabadi R, Yaghooti-Khorasani M, Ghazizadeh H, Ghaffarian-Zirak R, Nosrati-Tirkani A, Mohammadi-Bajgiran M, Rohban M, Sadabadi F, Rahimi HR, Ghalandari M, Ghaffari MS, Yousefi A, Pouresmaeili E, Besharatlou MR, Moohebati M, Ferns GA, Esmaily H, Ghayour-Mobarhan M. Dyslipidemia and cardiovascular disease risk among the MASHAD study population. Lipids Health Dis. 2020 Mar 16;19(1):42. doi: 10.1186/s12944-020-01204-y. PMID 32178672
- [Background] Firnhaber JM. Hyperlipidemia management: A calibrated approach. J Fam Pract. 2023 Apr;72(3):126-132. doi: 10.12788/jfp.0576. PMID 37075215
- [Background] Zhang X, Xing L, Jia X, Pang X, Xiang Q, Zhao X, Ma L, Liu Z, Hu K, Wang Z, Cui Y. Comparative Lipid-Lowering/Increasing Efficacy of 7 Statins in Patients with Dyslipidemia, Cardiovascular Diseases, or Diabetes Mellitus: Systematic Review and Network Meta-Analyses of 50 Randomized Controlled Trials. Cardiovasc Ther. 2020 Apr 23;2020:3987065. doi: 10.1155/2020/3987065. eCollection 2020. PMID 32411300
- [Background] Bharath G, Vishnuprabu DP, Preethi L, Nagappan AS, Dhianeshwaran Isravanya RT, Bhaskar LV, Swaminathan N, Munirajan AK. SLCO1B1 and ABCB1 variants synergistically influence the atorvastatin treatment response in South Indian coronary artery disease patients. Pharmacogenomics. 2022 Aug;23(12):683-694. doi: 10.2217/pgs-2022-0044. Epub 2022 Aug 15. PMID 35968761
- [Background] Na Nakorn C, Waisayarat J, Dejthevaporn C, Srisawasdi P, Wongwaisayawan S, Sukasem C. Genetic Variations and Frequencies of the Two Functional Single Nucleotide Polymorphisms of SLCO1B1 in the Thai Population. Front Pharmacol. 2020 Jun 5;11:728. doi: 10.3389/fphar.2020.00728. eCollection 2020. PMID 32581780
- [Background] Marin JJG, Serrano MA, Monte MJ, Sanchez-Martin A, Temprano AG, Briz O, Romero MR. Role of Genetic Variations in the Hepatic Handling of Drugs. Int J Mol Sci. 2020 Apr 20;21(8):2884. doi: 10.3390/ijms21082884. PMID 32326111
- [Background] Turongkaravee S, Jittikoon J, Lukkunaprasit T, Sangroongruangsri S, Chaikledkaew U, Thakkinstian A. A systematic review and meta-analysis of genotype-based and individualized data analysis of SLCO1B1 gene and statin-induced myopathy. Pharmacogenomics J. 2021 Jun;21(3):296-307. doi: 10.1038/s41397-021-00208-w. Epub 2021 Feb 19. PMID 33608664